CLINICAL TRIAL: NCT01433705
Title: Evaluation of the Normal Distribution of Rubidium-82(Rb-82), Nitrogen-13 (N-13)Ammonia, and Fluorine-18 Fluorodeoxyglucose (F-18FDG) in Normal Volunteers
Brief Title: Distribution of Rubidium-82, Nitrogen-13 Ammonia, and Fluorine-18 Fluorodeoxyglucose in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James R. Corbett, M.D., Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00016183
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Heart Disease
Keywords: heart; perfusion; glucose
MeSH Terms: conditions — Heart Diseases | interventions — regadenoson

STUDY DESIGN:
Intervention Model Description: Subjects will have a PET scan after IV administration of a radio-labelled tracer, Rb-82 and N-13 or injection of F-18 FDG
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rb-82 and N-13 ammonia Pet scans (Other): Rest and vasodilator stress Rb-82 images and N-13 ammonia images will be taken according to standard clinical imaging protocol. Each of these two imaging studies require the injection of Rb-82 and N-13 ammonia by intravenous administration (IV) in the patient's arm.
  Interventions: Other: Rb-82 Pet scans; Other: N-13 ammonia Pet scans; Drug: Regadenoson
- F-18 FDG Imaging and Rb-82 (Other): Volunteers not excluded by abnormal rest/stress imaging with Rb-82, will begin F-18 FDG protocol.
  Interventions: Other: Rb-82 Pet scans; Other: F-18 FDG Pet scans; Drug: Regadenoson
- F-18 FDG Imaging and N-13 ammonia (Other): Volunteers not excluded by abnormal rest/stress imaging with N-13 ammonia, will begin F-18 FDG protocol.
  Interventions: Other: F-18 FDG Pet scans; Other: N-13 ammonia Pet scans; Drug: Regadenoson

INTERVENTIONS:
Other: Rb-82 Pet scans — Intravenous administration of Rb-82. Images will be taken according to standard clinical imaging protocol and reviewed. Patient will be connected to an EKG machine to monitor the heart. Blood pressure will be monitored as well. For Rb-82 images, 40 mCi (millicuries are a measurement of radioactivity) will be used. Acquisition time for both rest and stress studies should take about 30 min.
  Arms: F-18 FDG Imaging and Rb-82; Rb-82 and N-13 ammonia Pet scans
Other: F-18 FDG Pet scans — Volunteers undergoing the F-18 FDG protocols will undergo: (1) glucose loading protocol for "viability protocol imaging" with the hyperinsulinemic euglycemic clamp according to standard procedures in our laboratory, and (2) "inflammation protocol imaging" using a high fat preparatory diet and three sub-therapeutic heparin doses (10 units / kg each) according to standard laboratory procedure. When metabolically prepared with the viability protocol and the inflammation protocol (two separate days), 10 mCi (millicuries) of F-18 FDG will be administered IV per FDG protocols, via heparin lock. 40-60 minutes after FDG injections PET imaging will be performed according to standard clinical imaging protocol.
  Arms: F-18 FDG Imaging and N-13 ammonia; F-18 FDG Imaging and Rb-82
Other: N-13 ammonia Pet scans — Intravenous administration of N-13. Images will be taken according to standard clinical imaging protocol and reviewed. Patient will be connected to an EKG machine to monitor the heart. Blood pressure will be monitored as well. For N-13 ammonia images, 20 mCi (millicuries) will be used. Acquisition time for both rest and stress studies should take about 30 min.
  Arms: F-18 FDG Imaging and N-13 ammonia; Rb-82 and N-13 ammonia Pet scans
Drug: Regadenoson — Regadenoson is used as a stressor; but not to study its effects.

SUMMARY:
Establish the normal distributions of Rb-82, N-13 ammonia, and F-18 FDG (radioactive tracers) in the heart using PET imaging. These tracers would be eventually used in evaluating the hearts of patients with heart disease.

Normal healthy volunteers will be carefully screened for this study. Subjects will be given IV administration of Rb-82 and N-13 to acquire rest/stress imaging. Normal subjects not excluded by any unexpected abnormality during the Rb-82 or N-13 rest/stress studies will undergo a glucose loading F-18 FDG imaging protocol, viability protocol using the hyperinsulinemic euglycemic clamp with simultaneous IV infusions of dextrose and insulin according to standard procedures in our laboratory.

These same subjects will have a F-18 FDG protocol after following a high fat, protein permitted, no carbohydrate diet for approximately 30 hours prior to F-18 FDG injection. The F-18 FDG radiotracer will be given through an IV.

DETAILED DESCRIPTION:
Cardiac rubidium-82(Rb-82)and N-13 ammonia heart perfusion (blood flow) studies and florine-18 fluorodeoxyglucose (F-18FDG) heart PET glucose metabolism studies are important tools for evaluating patients with coronary heart disease.

This includes patients with known or suspected heart disease and patients with congestive heart failure following myocardial infarction (heart attack) with indeterminant assessments of cardiac health from other types of imaging, such as SPECT perfusion imaging and echocardiography.

These studies help physicians plan potentially life saving procedures to re-establish coronary blood flow to living but severely compromised heart muscle. Rb-82 and N-13 ammonia studies can tell if there is reduced blood flow to the heart muscle either at rest or during stress.

FDG studies can tell whether there is any chance of a beneficial effect from coronary revascularization procedures, for example coronary angioplasties and stents or coronary artery bypass. Revascularization procedures in patients like these may be technically difficult, risky and costly.

Unfortunately the normal cardiac distributions of Rb-82, N-13 and ammonia, and F-18FDG for computer analysis of human studies are not well known and what is known is not widely available for clinical use. The latest imaging guidelines from the American Society of Nuclear Cardiology recommend that Rb-82, N-13 ammonia, and FDG cardiac studies be compared to normal distributions or patterns of these radiotracers in the heart developed from a series of normal individuals.

The purpose for these studies is to generate databases of normal Rb-82, N-13 ammonia, and F-18FDG cardiac distributions so that they can be used in the analysis of clinical patient studies at the University of Michigan Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal volunteers

Exclusion Criteria:

1. Prior participation in a study with significant radiation exposure
2. Significant radiation exposure for other reasons, example: routine medical care
3. Medical history of physical or treadmill exercise stress EKG evidence of heart or vascular disease.
4. Cardiac A-V conduction abnormalities
5. Diabetes Mellitus
6. Liver Disease
7. Kidney Disease
8. Other chronic debilitating illnesses ( Example: Rheumatoid Arthritis, Emphysema, Parkinson's Disease).
9. Tobacco use, hypertension, diabetes, family history of coronary artery disease before age 45 in males and 55 in females or other coronary risks factors of more than mild severity
10. Claustrophobia (fear of tight spaces)
11. Pregnancy
12. Inability to lay flat with your arms positioned next to your head for approximately 20 minutes.
13. Morbid Obesity
14. Asthma
15. Breasts Implants
16. Use of anabolic steroids
17. Use of recreational drugs

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
analysis of healthy cardiac distribution of Rb-82, N-13 ammonia, and F-18 FDG. | approximately 4 to 10 hours
  Normal healthy volunteers will undergo PET imaging during vasodilator pharmacologic stress with regadenoson and at rest with Rb-82 and or N-13 ammonia and or at rest with F-18FDG. Participants will have either rest and stress Rb-82 and rest and stress N-13 ammonia or one of these stress tests and F-18 FDG imaging.

CONTACTS AND LOCATIONS:
Overall Officials: James R. Corbett, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No